CLINICAL TRIAL: NCT05033834
Title: Covid-19 Infection in Partially and Fully Vaccinated Cases: Cohort Study
Brief Title: Covid-19 Infection in After Vaccination
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aliae AR Mohamed Hussein, Professor of Pulmonology, Assiut University
Other Study IDs: Assiut-breakthrough covid-19
Record Dates: First submitted 2021-09-02; First posted 2021-09-05 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Covid19
Keywords: COVID-19; COVID-19 vaccination; Post vaccination infection; breakthrough COVID-19; Partially vaccinated; Fully vaccinated
MeSH Terms: conditions — COVID-19; COVID-19 breakthrough infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: People received any registered COVID-19 vaccination
  Interventions: Other: covid-19 vaccines registered in Egypt
- Group B: People developed COVID-19 infection after partial or full vaccination with any registered COVID-19 vaccine
  Interventions: Other: covid-19 vaccines registered in Egypt

INTERVENTIONS:
Other: covid-19 vaccines registered in Egypt — Astra Zeneka vaccine, Sinopharm vaccine, Sinovac vaccine, Jonson and Jonson vaccine, Spotnic V vaccine

SUMMARY:
Coronavirus disease 2019 (COVID-19), caused by severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), was first identified in Wuhan, China. It rapidly spread, resulting a global pandemic in March 2020. Globally, till 27 August 2021, there have been 214,468,601 confirmed cases of COVID-19, including 4,470,969 deaths, reported to WHO.

With the absence of curative treatment for COVID-19 infection the development of safe and effective vaccines is critical to ending the COVID-19 pandemic. The Pfizer/BioNtech Comirnaty vaccine was listed for WHO Emergency Use Listing (EUL) on 31 December 2020. The SII/Covishield and AstraZeneca/AZD1222 vaccines (developed by AstraZeneca/Oxford and manufactured by the State Institute of India and SK Bio respectively) were given EUL on 16 February. The Janssen/Ad26.COV 2.S developed by Johnson & Johnson, was listed for EUL on 12 March 2021. The Moderna COVID-19 vaccine (mRNA 1273) was listed for EUL on 30 April 2021 and the Sinopharm COVID-19 vaccine was listed for EUL on 7 May 2021. The Sinopharm vaccine is produced by Beijing Bio-Institute of Biological Products Co Ltd, subsidiary of China National Biotec Group (CNBG). The Sinovac-CoronaVac was listed for EUL on 1 June 2021. As of 25 August 2021, a total of 4,953,887,422 vaccine doses have been administered. In large, randomized-controlled trials, vaccines were found to be safe and efficacious in preventing symptomatic, laboratory-confirmed COVID-19.

However, a small percentage of fully vaccinated persons will develop symptomatic or asymptomatic infections with SARS-CoV-2, the virus that causes COVID-19. A vaccine breakthrough infection is defined as the detection of SARS-CoV-2 RNA or antigen in a respiratory specimen collected from a person ≥14 days after receipt of all recommended doses of an FDA-authorized COVID-19 vaccine. A total of 10,262 SARS-CoV-2 vaccine breakthrough infections had been reported from 46 U.S. states and territories as of April 30, 2021. Among these cases, 6,446 (63%) occurred in females, and the median patient age was 58 years (interquartile range = 40-74 years). Based on preliminary data, 2,725 (27%) vaccine breakthrough infections were asymptomatic, 995 (10%) patients were known to be hospitalized, and 160 (2%) patients died.

ELIGIBILITY:
Inclusion Criteria:

* • Patients 18 years old and above of both genders.

  * Received at least one dose of COVID-19 registered vaccines.
  * Diagnosed COVID-19 positive after vaccination by real time PCR (confirmed case) or combined clinical and radiological diagnosis (possible case).

Exclusion Criteria:

• Children less than 18 years.

* Cases non vaccinated with COVID-19 registered vaccine

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Group A: people receive vaccination at the study period will be followed by phone calls or email for any new infection. Group B: patients who will be confirmed to have recent COVID-19 infection who visit outpatient clinic or admit to ward or ICU of Assiut University hospital at study period.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
assess the prevalence of COVID-19 infection after vaccination | one year
  number of cases with covid-19 after vaccination

SECONDARY OUTCOMES:
evaluate the severity of infection after vaccination | 2 weeks
  severity of covid-19 infection in partially and fully vaccinated cases
Predict possible risk factors of post vaccination infection | one year
  adherence to protective measures

CONTACTS AND LOCATIONS:
Locations (3):
- Egypt (3):
  - AssiutU, Asyut
  - Pulmonology Departments, Asyut
  - Aliae AR Mohamed-Hussein, Asyut

IPD SHARING:
Plan to Share IPD: Undecided
upon reasonable request